CLINICAL TRIAL: NCT05517083
Title: Feasibility of Intratumoral Washing Fluid for Detecting EGFR Mutations in Advanced Non-small Cell Lung Cancer
Brief Title: Feasibility of Intratumoral Washing Fluid for Detecting EGFR Mutations in Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2204-006-113
Record Dates: First submitted 2022-07-30; First posted 2022-08-26 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Non Small Cell Lung Cancer; EGFR Gene Mutation
Keywords: Carcinoma, Non-Small-Cell Lung; EGFR Genes; Bronchoscopy; Liquid biopsy; T790M
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrathin bronchoscopy with intratumoral washing (Experimental): Each subject with NSCLC will undergo bronchooscopic procedure for EGFR mutation (including T790M positivity) evaluation.
  Interventions: Diagnostic Test: Ultarthin bronchoscopy with intratumoral washing

INTERVENTIONS:
Diagnostic Test: Ultarthin bronchoscopy with intratumoral washing — Each subject with NSCLC will undergo bronchooscopic procedure. First, ultrathin bronchoscope is inserted and placed within tumor under radial EBUS, virtual bronchoscopic navigation, and fluoroscopy guidance. Then, intratumoral washing is performed. Subsequently, transbronchial lung biopsy is performed under radial EBUS, virtual bronchoscopic navigation, and fluoroscopy guidance.

SUMMARY:
The purpose of this study is to evaluate the relevance of intratumoral washing for detection of EGFR mutation (including T790M positivity).

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label study to assess evaluate the relevance of intratumoral washing by ultrathin bronchoscopy (outer diameter; 3mm) for detection of EGFR mutation (including T790M positivity) using cobas real-time PCR and droplet digital PCR (DDPCR) in patients with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Obtained written informed consent
* Patients diagnosed with NSCLC by histology or cytology and inoperable stage IV at the time of study enrollment
* Patients with the following EGFR gene mutations: E19Del, L858R alone or concurrent rare EGFR gene mutations (T790M, G719X, exon 20 insertion, S768I)
* Patients previously treated with EGFR-TKIs such as gefitinib, erlotinib, afatinib, dacomitinib as first line therapy
* Patients who had shown clinical benefits (CR, PR, SD) from EGFR-TKIs and had been confirmed PD on those therapy according to RECIST v 1.1.
* Patients who underwent liquid biopsy (plasma) for EGFR mutation at the time of PD on EGFR-TKIs
* Patients who plan to undergo tissue biopsy for EGFR mutation at the time of PD on EGFR-TKIs

Exclusion Criteria:

* Patients who withdraw informed consent
* Patients who are unable to undergo liquid biopsy (plasma) and tissue biopsy for EGFR mutation based on the investigator's judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The DNA and EGFR mutation (including T790M positivity) detection rate in intratumoral washing fluid | through study completion, an average of 1 year
  Defined as the number of DNA and EGFR mutation (including T790M positivity) detection divided by the total attempts of intratumoral washing by ultrathin bronchoscopy.

SECONDARY OUTCOMES:
The concordance rate of EGFR mutation (including T790M positivity) detection rate among intratumoral washing fluid, plasma, and tissue | through study completion, an average of 1 year
  The concordance rate of EGFR mutation (including T790M positivity) detection rate in intratumoral washing fluid, compared with plasma and tissue (gold standard).
The EGFR mutation (including T790M positivity) sensitivity and specificity in intratumoral washing fluid | through study completion, an average of 1 year
  The sensitivity and specificity of EGFR mutation (including T790M positivity) in intratumoral washing fluid compared with tissue (gold standard).
Objective response rate | through study completion, an average of 1 year
  Objective response rate (ORR) including rate of complete response (CR) and partial response (PR) based on RECIST 1.1.
Disease control rate | through study completion, an average of 1 year
  Disease control rate (DCR) including rate of CR, PR and stable disease (SD) based on RECIST 1.1.
Progression-free survival | through study completion, an average of 1 year
  Progression-free survival (PFS) the time from first dose of the study drug until the date of progressive disease (PD) based on RECIST 1.1 or death by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Hyun Kim, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University hospital, Busan, South Korea